CLINICAL TRIAL: NCT04845087
Title: Pilot Study for the Management of Peri-implant Mucositis With Ozone Water Jet: a Randomized Clinical Trial.
Brief Title: Management of Peri-implant Mucositis With Ozone Water Jet: a Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Research Resident, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-AQUALAB
Record Dates: First submitted 2021-04-13; First posted 2021-04-14 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Peri-implant Mucositis
Keywords: ozonized water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial Group (Experimental): Patients from this group will receive treatment with ozonized water.
  Interventions: Other: Ozonized water
- Placebo Group (Placebo Comparator): Patients from this group will receive placebo with water.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Ozonized water — Irrigation of dental implants with ozonized water
  Arms: Trial Group
Other: Placebo — Irrigation of dental implants with water
  Arms: Placebo Group

SUMMARY:
The aim of this study is to assess if ozonized water can be used for the treatment of peri-implant mucositis in patients with dental implants.

Patients willl undergo professional dental hygiene also with the use of glycine powders, then they will be randomly divided into two groups:

* Trial Group: irrigation of peri-implant periodontium with mucositis with ozonized water.
* Placebo Group: irrigation of peri-implant periodontium with mucositis with water.

Periodontal indices will be recorded at the baseline, after 1 and 2 months. After 1 and 2 months, only glycine powders will be performed, together with ozonized water or water irrigation and the collection of periodontal indices.

DETAILED DESCRIPTION:
The aim of this study is to assess if ozonized water can be used for the treatment of peri-implant mucositis in patients with dental implants.

Patients who respond to eligibility criteria and that will sign the informed consent will undergo a professional oral hygiene procedure.

Patients willl undergo professional dental hygiene also with the use of glycine powders. Then, glycine powders air-flow will be administered. Then they will be randomly divided into two groups:

* Trial Group: irrigation of peri-implant periodontium with mucositis with ozonized water.
* Placebo Group: irrigation of peri-implant periodontium with mucositis with water.

Periodontal indices will be recorded at the baseline, after 1 and 2 months. After 1 and 2 months, only glycine powder will be performed, together with ozonized water/water irrigation and the collection of periodontal indices.

ELIGIBILITY:
Inclusion Criteria:

* Presence of one or more dental implants
* Presence of peri-implant mucositis at least at one implant
* Bleeding Score > 0

Exclusion Criteria:

* Patents without dental implants
* Presence of systemic diseases
* Patients with cardiac pacemaker

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-04-24 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Change in PPD - Probing Depth | Baseline, 1 and 2 months.
  Evaluation (in mm) of the depth of the gingival sulcus, through a millimeter periodontal probe; it is detected from the gingival margin to the bottom of the gingival sulcus of the peri-implant pocket, evaluated at 6 sites.
Change in BOP - Bleeding on Probing (percentage) | Baseline, 1 and 2 months.
  Site-specific assessment of the presence or absence of gum bleeding after the insertion of the periodontal probe for the detection of PD, detected on 6 sites.
Change in BS - Bleeding Score | Baseline, 1 and 2 months.
  Scoring criteria:
  * 0: no bleeding;
  * 1: punctiform bleeding in the site of probing;
  * 2: bleeding within the gingival border;
  * 3: bleeding outside the gingival border.
Change in PI - Plaque Index (percentage) | Baseline, 1 and 2 months.
  Site-specific assessment of the presence or visible plaque detected on 4 sites with a disclosing tables.
  Percentage of sites with plaque determines the PI%.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD., Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator.